CLINICAL TRIAL: NCT04939584
Title: A Clinical Feasibility Study to Evaluate Patient Perception of MPT
Brief Title: Patient Perception of MultiPulse Therapy™ (MPT™)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor ceased operations
Sponsor: Cardialen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL008
Record Dates: First submitted 2021-06-10; First posted 2021-06-25 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A prospective non-randomized feasibility study involving acute evaluation of the perception and acceptance of MPT as a therapy to stop episodes of AF in subjects having a history of AF during clinically indicated acute electrophysiology procedures including AF ablation, SVT ablation or diagnostic EP procedures (indicated procedure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): The study will be conducted using the venous cannulations that are standard of care for the indicated procedure. Additional access points may be necessary if access to coronary sinus is difficult from existing femoral venous cannulations. Sterile study leads or EP catheters will be temporarily placed into the RA, CS, and RV (for R-wave sensing using intracardiac electrograms - optional) which will be connected to the investigational device (CESS).
  Up to two MPTs will be delivered and subject responses following each MPT regarding perception and acceptability of MPT to treat AF will be obtained. MPT voltages will not exceed 100V.
  Interventions: Device: MultiPulse Therapy

INTERVENTIONS:
Device: MultiPulse Therapy — Electrical Stimulation

SUMMARY:
Assess the subject acceptance of MPT, using therapy parameters that have been shown to be effective in terminating episodes of atrial fibrillation.

DETAILED DESCRIPTION:
A prospective non-randomized feasibility study involving acute testing of MPT in subjects having a history of AF during clinically indicated acute electrophysiology procedures including AF ablation, SVT ablation or diagnostic EP procedures (indicated procedure). The primary outcome of the study is the subject response to questions regarding perception and acceptability following MPT delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 80 years of age
2. Willing and able to comply with the study protocol, provide a written informed consent
3. History of Atrial Fibrillation in past 12 months
4. Indicated to undergo an acute electrophysiology procedure allowing for conscious participation in the clinical study
5. Current treatment and compliance with standard anticoagulation regimen, including uninterrupted OAC, with acceptable coagulation status, as determined by the Principal Investigator

Study stage dependent: Stage 1:

6a. History of DC-Cardioversion in past 12 months: With or Without

7b. AFEQT Score: <=89

Study stage dependent: Stage 2 (based on results from study stage 1):

6a: History of DC-Cardioversion in past 12 months: Potential emphasis on patients with history of DCCV

7b. AFEQT Score: Potential emphasis on patients with AFEQT <= 58

Exclusion Criteria:

1. Life expectancy of 1 year or less
2. AF due to reversible causes (e.g., hyperthyroidism, valve disease)
3. Hx of fibromyalgia or any other evidence of wide-spread pain
4. Any current pain condition that could be confused with pain or discomfort associated with MPT
5. >1 current well-defined pain condition (e.g., migraine, joint OA, painful diabetic neuropathy)
6. Use of any opioid analgesic (including tramadol) within 3 months of screening
7. Spielberger's STAI-AD-Trait > 75
8. AFEQT: Section 1: "I was never aware of having atrial fibrillation" is checked
9. Allergy or contraindication to anticoagulation therapy
10. Presence of intracardiac thrombus (confirmed with cardiac imaging)
11. Existing Left Atrial Appendage closure device
12. LVEF<20%
13. NYHA Class IV heart failure at the time of enrollment
14. History of embolic stroke, Transient Ischemic Attack (TIA) or other thromboembolic event within the preceding 3 months.
15. Known hyper-coagulable state that increases risk of thrombus
16. History of myocardial infarction or coronary revascularization within the preceding 3 months.
17. History of sustained ventricular arrhythmia or cardiac arrest
18. Presence of chronically implanted lead in the CS
19. Presence of ventricular assist device, including intra-aortic balloon pump
20. Documented bradycardia (<40 BPM) at the time of the study
21. Morbid obesity: BMI>39 kg/m2
22. Presence of any prosthetic cardiac valve
23. History of significant tricuspid valvular disease requiring surgery
24. Moderate to severe mitral valve regurgitation (>40% regurgitation fraction)
25. Cognitive or mental health status that would interfere with study participation and proper informed consent
26. Cardiovascular anatomical defects that would complicate placement of the stimulation leads required by the protocol, including congenital heart disease and cardiac vein anomalies per the Investigator's discretion
27. Pregnancy confirmed by test within 7 days of procedure.
28. Inability to pass catheters to heart due to vascular limitations
29. Cardiovascular surgery or intervention within 1 month prior to enrollment or planned for up to 1 month after enrollment (other than the planned treatment procedure)
30. Active endocarditis
31. History of hemodynamic compromise due to valvular heart disease
32. Unstable CAD as determined by the investigator
33. Severe proximal three-vessel or left main coronary artery disease without revascularization as determined by the investigator
34. History of Hypertrophic Cardiomyopathy, Arrhythmogenic Right Ventricular Dysplasia, Congenital Heart Anomaly, Cardiac Amyloidosis or Cardiac Sarcoidosis
35. Any other medical condition which may affect the outcome of this study or safety of the subject as determined by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Therapy acceptance as measured by a subject question administered immediately following MPT delivery | Immediately following MPT delivery
  Question: "Now I want you to think about your experiences with Atrial Fibrillation. Think about how it makes you feel, your daily life while in atrial fibrillation and your experience with in-clinic treatments for atrial fibrillation. If you could use the stimulation you just felt at home and under your control, would you use this stimulation therapy to stop your atrial fibrillation? Please answer yes or no."
Subject perception of MPT as measured by a pain scale administered immediately following MPT delivery | Immediately following MPT delivery
  Question: "Please rate any pain you experienced at the time of the stimulus, was it: No pain, mild pain, moderate pain, severe pain, the worst possible pain imaginable."?

SECONDARY OUTCOMES:
Safety determined from summary report of Adverse Events | Through 30 days post-intervention
  Adverse Event frequency by Adverse Event type

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St. Andrew's Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No